#### CLINICAL STUDY PROTOCOL

# A 6-MONTH, MULTICENTER, PHASE 3, OPEN-LABEL EXTENSION SAFETY STUDY OF OTO-104 GIVEN AT 3-MONTH INTERVALS BY INTRATYMPANIC INJECTION IN SUBJECTS WITH UNILATERAL MENIERE'S DISEASE

**Protocol Number: 104-201509** 

Sponsor Contact:

Medical Monitor:

Version: 2.0

Date of Protocol: 22 February 2016

Proprietary Notice The concepts and information contained in this document or generated

during the study are considered proprietary and may not be disclosed in whole or in part without the expressed, written consent of Otonomy,

Inc.

#### CONFIDENTIALITY STATEMENT

The information in this document contains trade secrets and commercial information that are privileged or confidential and may not be disclosed unless such disclosure is required by applicable laws and regulations. In any event, persons to whom the information is disclosed must be informed that the information is privileged or confidential and may not be further disclosed by them. These restrictions on disclosure will apply equally to all future information supplied to you which is indicated as privileged or confidential.

A 6-MONTH, MULTICENTER, PHASE 3, OPEN-LABEL EXTENSION SAFETY STUDY OF OTO-104 GIVEN AT 3-MONTH INTERVALS BY INTRATYMPANIC INJECTION IN SUBJECTS WITH UNILATERAL MENIERE'S DISEASE

## APPROVED BY:



#### MEDICAL MONITOR:

I acknowledge that I have read and understood this protocol.



# TABLE OF CONTENTS

| TITLE I | PAGE | 1 |
|---------|---------------------------------------------------------------|----|
| PROTO | COL AMENDMENT, VERSION 2.0 | 7 |
| SPONS | OR CONTACT INFORMATION | 8 |
| INVEST | TIGATOR AGREEMENT | 9 |
| ABBRE | VIATIONS | 10 |
| SYNOP | SIS | 11 |
| 1. | BACKGROUND | 15 |
| 1.1. | Rationale for Safety Study | 16 |
| 2. | OBJECTIVES | 16 |
| 3. | OVERVIEW OF STUDY DESIGN | 16 |
| 4. | STUDY POPULATION | 17 |
| 4.1. | General Considerations | 17 |
| 4.2. | Inclusion Criteria | 17 |
| 4.3. | Exclusion Criteria | 17 |
| 5. | RANDOMIZATION AND BLINDING | 18 |
| 5.1. | Enrollment Procedures | 18 |
| 5.1.1. | Assignment of Subject Identification Numbers | 18 |
| 6. | DOSAGE AND ADMINISTRATION | 18 |
| 6.1. | Study Drug Administration | 18 |
| 6.2. | Compliance | 19 |
| 7. | PRIOR, CONCOMITANT, AND SUBSEQUENT THERAPY | 19 |
| 7.1. | Proscribed Therapy or Procedures During the Study Period | 19 |
| 7.2. | Symptomatic Relief Medications | 20 |
| 8. | STUDY EVALUATIONS | 20 |
| 8.1. | Study Procedures by Visit | 20 |
| 8.1.1. | Visit 1: Day 1 (Screening/Baseline/Dose No. 1) | 20 |
| 8.1.2. | Visit 2: Month 3 (± 2 weeks) (Follow Up and Dose No. 2) | 20 |
| 8.1.3. | Visit 3: Month 6 (± 2 weeks) (End of Study/Early Termination) | 21 |
| 8.1.4. | Unscheduled Visit | 21 |
| 8.2. | Safety Evaluations | 22 |
| 8.2.1. | Vital Sign, Height and Weight Measurements | 22 |

| 8.2.2. | Urine Pregnancy Test | 22 |
|---|---|---|
| 8.2.3. | Tympanometry | 22 |
| 8.2.4. | Audio grams | 22 |
| 8.2.5. | Otoscopy | 23 |
| 8.2.6. | C-SSRS Assessment | 23 |
| 8.3. | Additional Evaluations | 23 |
| 8.3.1. | Meniere's Symptom Questionnaire | 23 |
| 9. | ADVERSE EVENT (AE) REPORTING | 24 |
| 9.1. | Adverse Event Classification Definitions | 24 |
| 9.1.1. | Assessment of Severity | 25 |
| 9.1.2. | Assessment of Causality | 25 |
| 9.1.3. | Follow up of Adverse Events | 26 |
| 9.2. | Monitoring of Adverse Events | 26 |
| 9.2.1. | All Adverse Events | 26 |
| 9.2.2. | Serious Adverse Events | 27 |
| 9.2.3. | Pregnancies | 27 |
| 9.3. | Contacting Sponsor Regarding Safety | 27 |
| 10. | SUBJECT COMPLETION | 28 |
| 10.1. | Completion | 28 |
| 10.2. | Withdrawal | 28 |
| 10.2.1. | Handling of Withdrawals | 28 |
| 10.2.2. | Replacements | 29 |
| 11. | STATISTICAL METHODS | 29 |
| 11.1. | Sample Size | 29 |
| 11.2. | Analysis Sets | 29 |
| 11.3. | Description of Subgroups to be Analyzed | 29 |
| 11.4. | Subject Demographics, Baseline Disease Status, and Disposition | 29 |
| 11.5. | Efficacy Evaluations | 29 |
| 11.6. | General Analytic Methods | 30 |
| 11.7. | Safety Evaluations | 30 |
| 11.7.1. | Adverse Events | 30 |
| 11.7.2. | Vital Signs | 30 |
| 11.7.3. | Otoscopic Examinations | 30 |

| 11.7.4. | Audiometry Assessments | 31 |
|---|---|---|
| 11.7.5. | Tympano metry | 31 |
| 11.7.6. | Concomitant Medications | 31 |
| 11.7.7. | C-SSRS | 31 |
| 11.7.7.1. | C-SSRS: Baseline Version | 31 |
| 11.7.7.2. | C-SSRS: Since Last Visit Version | 31 |
| 11.8. | Other Evaluations | 32 |
| 11.8.1. | Meniere's Symptom Questionnaire | 32 |
| 11.9. | Handling of Missing Data, Subject Withdrawals, and Treatment Failures | 32 |
| 11.10. | Interim Analyses | 32 |
| 12. | STUDY DRUG INFORMATION | 32 |
| 12.1. | Physical Description of Study Drug(s) | 32 |
| 12.2. | Directions for Use | 33 |
| 12.3. | Packaging and Labeling | 33 |
| 12.3.1. | Packaging | 33 |
| 12.3.2. | Labels and Labeling Instructions | 33 |
| 12.4. | Management of Clinical Supplies | 33 |
| 12.4.1. | Storage of Kits | 33 |
| 12.5. | Drug Accountability | 33 |
| 13. | ETHICAL ASPECTS | 34 |
| 13.1. | Investigator Responsibilities | 34 |
| 13.2. | Institutional Review Board (IRB) | 34 |
| 13.3. | Informed Consent | 34 |
| 14. | ADMINISTRATIVE REQUIREMENTS | 35 |
| 14.1. | Protocol Modifications | 35 |
| 14.2. | Regulatory Documentation | 35 |
| 14.3. | Subject Identification Register | 36 |
| 14.4. | Record Retention | 36 |
| 14.5. | Electronic Case Report Form. | 36 |
| 14.6. | Termination | 37 |
| 14.7. | Data and Safety Monitoring Plan | 37 |
| 14.8. | Monitoring | 37 |
| 14.9. | Data Quality Assurance | 38 |

| 14.10. | On-Site Audits | 38 |
|--------|-------------------------------------|----|
| 14.11. | Use of Information and Publication. | 38 |
| 15. | LIST OF REFERENCES | 40 |

# PROTOCOL AMENDMENT, VERSION 2.0

This protocol amendment serves to make the following changes.

| Item<br>No. | Change | Section and Page Number |
|---|---|---|
| 1 | Updated date and version of protocol. | Title page, pg. 1 Footer, every page |
| 2 | Safety reporting changed to | Sponsor Contact Information, pg. 8 Section 9.3 Contacting Sponsor Regarding Safety, pg. 27 |
| 3 | Added additional exclusion criteria to hypersensitivity to dexamethasone or any of the OTO-104 excipients. | Synopsis, pg. 12<br>Section 4.3 Exclusion Criteria, pg. 18 |
| 4 | Added 3-digit identification number to the subject number to indicate which study the subject was previously enrolled in. | Section 5.1.1 Assignment of Subject<br>Identification Numbers, pg. 18 |
| 5 | Corrected visit numbers. | Section 6.2 Compliance, pg. 19 |

# **SPONSOR CONTACT INFORMATION**

# Medical Monitor: Name Title Office Phone Number Mobile Phone Number E-Mail Other Appropriate Trial Contact Personnel: Name Title Office Phone Number Mobile Phone Number E-Mail Safety Email:

If any sponsor contact information needs to be changed during the course of the study, this will be done by the sponsor, with written notification to the investigator, and will not require a protocol amendment.

#### INVESTIGATOR AGREEMENT

I have read this protocol and agree that it contains all necessary details for carrying out this study. I will conduct the study as outlined herein and will complete the study within the time designated and will abide by all obligations stated on the Form FDA 1572 and other local regulatory authority required document(s).

I will provide copies of the protocol and all pertinent information to all individuals responsible to me who assist in the conduct of this study. I will discuss this material with them to ensure they are fully informed regarding the drug and the conduct of the study.

I will use only the informed consent form approved by the sponsor or its representative and approved by the Institutional Review Board (IRB) responsible for this study and will fulfill all responsibilities for submitting pertinent information to the IRB responsible for this study. I will assure that each subject enrolled into the trial, or legally authorized representative, reads, understands, and signs the appropriate version of the informed consent. I agree that the sponsor or its representatives shall have access to any original source documents to verify data captured for this clinical trial.

I further agree not to originate or use the name of the Otonomy, Inc. and/or OTO-104, or any of its employees, in any publicity, news release or other public announcement, written or oral, whether to the public, press or otherwise, relating to this protocol, to any amendment hereto, or to the performance hereunder, without the prior written consent of Otonomy, Inc.

| Investigator's Signature | Date |
|-----------------------------------------|------|
| Name of Investigator (typed or printed) | |
| Institution Name | |

## **ABBREVIATIONS**

Abbreviation Explanation

AAO-HNS American Academy of Otolaryngology - Head and Neck Surgery

AE Adverse Event

BCA Bone Conduction Average

C Celsius

CRF/eCRF Case Report Form/electronic Case Report Form

CRO Contract Research Organization

C-SSRS Columbia-Suicide Severity Rating Scale

dB Decibel

EDC Electronic Data Capture System

F Fahrenheit
FAX Facsimile

FDA Food and Drug Administration

GCP Good Clinical Practice

HIPAA Health Insurance Portability and Accountability Act

Hz Hertz

ICH International Conference on Harmonization

IRB Institutional Review Board

IT Intratympanic

MedDRA Medical Dictionary for Regulatory Activities

mL Milliliter
mg Milligram
mm Millimeter

OTO-104 Investigational Product
PTA Pure Tone Average
SAE Serious Adverse Event
SAP Statistical Analysis Plan

SOC System Organ Class

TEAE Treatment Emergent Adverse Event

#### **SYNOPSIS**

NAME OF SPONSOR/COMPANY: Otonomy, Inc.

NAME OF INVESTIGATIONAL PRODUCT: OTO-104

NAME OF ACTIVE INGREDIENT: Dexamethasone

**Title of Study:** A 6-month, multicenter, Phase 3, open-label extension safety study of OTO-104 given at 3-month intervals by intratympanic injection in subjects with unilateral Meniere's disease.

Study Center(s): This study will be conducted at approximately 60-70 sites in the United States.

Studied Period: 18 months Phase of Development: Phase 3

#### Study Design:

This is a 6-month, multicenter, Phase 3, open-label extension safety study in subjects with unilateral Meniere's disease. Subjects will receive 1 intratympanic (IT) injection of 12 mg OTO-104 at 3-month intervals for a total of 2 injections. Safety data to be collected include adverse events, concomitant medications, otoscopy, vital signs, audiology, tympanometry, Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire and a Meniere's disease symptom questionnaire.

#### Objective:

The objective is to assess the safety of repeat IT injections of 12 mg OTO-104 at 3-month intervals in an open-label study.

## Methodology:

The duration of the study for each subject will be 6 months.

Once subjects meet all eligibility criteria, they will be enrolled and may receive up to 2 IT injections of OTO-104 at 3-month intervals. All subjects will remain on standard of care treatment for unilateral Meniere's disease. Subjects will return to the study sites at Month 3 for safety assessments and another IT injection of OTO-104. Safety assessments will be completed at the end of the study (Month 6) or upon early withdrawal from the study.

#### Number of Subjects:

Up to 300 subjects will be enrolled.

#### Diagnosis and Main Criteria for Inclusion:

Subjects enrolled in the study will have unilateral Meniere's disease as outlined by the American Academy of Otolaryngology - Head and Neck Surgery (AAO-HNS) Committee on Hearing and Equilibrium in 1995 (Committee on Hearing and Equilibrium, 1995).

To be eligible for this study, each of the following criteria must be satisfied with a "YES" answer (unless not applicable):

- 1. Subject is a male or female aged 18 years or older.
- 2. Subject has completed the Phase 2b (104-201102) or Phase 3 (104-201506) clinical study.
- 3. Female subjects of childbearing potential [i.e., not surgically sterile and/or not postmenopausal (≥12 months since last menstrual period and 45 years of age or older)] must have

a negative urine pregnancy test before enrollment. Women of childbearing potential who are not abstinent from sex with male partners may be entered into the study if they are using and willing to continue to use highly effective or "double barrier" contraceptive precautions for the duration of the study (e.g., oral contraceptives, contraceptive implant or injection, intrauterine device, or "double barrier" methods including condom with diaphragm, male condom with cervical cap, male condom with spermicide, or diaphragm and spermicide).

- 4. Subject is willing to comply with the protocol and attend all study visits.
- Subject is able to provide written informed consent, including agreement to privacy language either within the informed consent or in ancillary documents compliant with Health Insurance Portability and Accountability Act (HIPAA), before the initiation of any study-related procedures.

#### Diagnosis and Main Criteria for Exclusion:

To be eligible for this study, each of the following criteria must be satisfied with a "NO" answer: (unless not applicable):

- 1. Subject has an infection in the ear, sinuses, or upper respiratory system.
- 2. Subject is pregnant or lactating.
- 3. Subject has a history of immunodeficiency disease.
- 4. Subject has active or recent (<1 month prior to screening) middle ear disease, including but not limited to: chronic otitis media, acute otitis media, middle ear effisions, middle ear atelectasis, or cholesteatoma.
- 5. Subject has an abnormality of the tympanic membrane in the affected ear that would increase the risk associated with intratympanic injection including but not limited to a monomeric, atelectatic or atrophic tympanic membrane.
- 6. Subject has a history of tympanostomy tubes that includes evidence of perforation or lack of closure.
- 7. Subject has a history of previous endolymphatic sac surgery.
- 8. Subject has a history of previous use of intratympanic gentamic in the affected ear.
- 9. Subject has history of drop attacks.
- 10. Subject has used systemic steroids within 1 month prior to Visit 1.
- 11. Subject has had intratympanic steroids within 1 month prior to Visit 1.
- 12. Subject has experienced an adverse reaction to intratympanic injection of steroids.
- 13. Subject has a hypersensitivity to dexamethasone or any of the excipients in OTO-104.
- 14. Subject has any other clinically significant illness or medical condition that, in the investigator's and the medical monitor's opinion, would prohibit the subject from participating in the study.
- 15. Subject has participated in a clinical trial within 30 days of Visit 1, not including the OTO-104 Phase 3 study (104-201506).

#### Criteria for Evaluation:

#### Safety Evaluations:

Key safety assessments include:

- Adverse events
- Audiometry assessments
- Tympanometry
- Local tolerability (otoscopic examinations)
- Vital sign measurements
- Columbia-Suicide Severity Rating Scale (C-SSRS): Baseline and Since Last Visit versions

#### Other Evaluations:

• Meniere's symptom questionnaire

#### Statistical Methods:

This is an open label safety study with one treatment group. All statistical analyses will be descriptive in nature.

## Investigational Product, Dosage and Mode of Administration:

OTO-104 12 mg, single, intratympanic injection, 0.2 mL

#### **Duration of Treatment:**

Single IT injection given at Day 1 and Month 3

# Reference Therapy, Dosage and Mode of Administration:

None

Time and Events Schedule: See Table 1.

Table 1: **Time and Events Table** 

| | Screening/<br>Baseline/Dose<br>No. 1 | Follow-up/ Dose<br>No. 2 | End-of-Study/<br>Early Term. | Unscheduled<br>Visit |
|---|---|---|---|---|
| | Visit 1 | Visit 2 | Visit 3 <sup>2</sup> | Unscheduled |
| Procedure | Day 1 | Month 3<br>(± 2 weeks) | Month 6<br>(± 2 weeks) | N/A |
| Informed consent (including privacy documents) | X | | | |
| Eligibility criteria | X | | | |
| Medical history <sup>3</sup> | X | | | |
| Concomitant medications | X | X | X | X |
| Vital sign measurements <sup>4</sup> | X | X | X | X |
| Height and weight measurements | X | | x <sup>5</sup> | |
| Urine Pregnancy test <sup>6</sup> | X | X | X | |
| Tympanometry | X | X | X | X as indicated |
| Audiometry | X | X | X | X as indicated |
| Otoscopy | X | X | X | X |
| C-SSRS assessment <sup>7</sup> | X | X | X | X |
| Meniere's symptom<br>questionnaire | X | X | X | |
| Administer study drug | X | X | | |
| Adverse event monitoring | X | X | X | X |

<sup>&</sup>lt;sup>1</sup> Visit 1 may also be the last study visit for 104-201506.

<sup>&</sup>lt;sup>2</sup> Procedures scheduled for Visit 3 will be performed at the end of the follow-up period (± 2 weeks) or upon early discontinuation from the study.

<sup>3</sup> Medical history to include information on demographics.

<sup>&</sup>lt;sup>4</sup> Vital sign measurements include blood pressure and pulse rate.

<sup>&</sup>lt;sup>5</sup> Only weight will be taken at Study Visit 3.

<sup>&</sup>lt;sup>6</sup> Female subjects of childbearing potential will have a urine pregnancy test via dipstick at every scheduled visit. On Visit 1 and 2, the pregnancy test must be completed and confirmed negative prior to dosing. If a subject is found to be pregnant after dosing with OTO-104, they will complete the follow-up period but will not be dosed further

<sup>&</sup>lt;sup>7</sup> At Visit 1, the Since Last Visit version of the C-SSRS will be used for subjects enrolling from Study 104-201506 while the Baseline version will be used for all subjects enrolling from Study 104-201102. The Since Last Visit version of the C-SSRS will be used at all subsequent visits.

#### 1. BACKGROUND

Meniere's disease is an idiopathic syndrome of endolymphatic hydrops (Committee on Hearing and Equilibrium, 1995). It is associated with a distinct pattern of clinical symptoms comprised of vertigo, hearing loss, timitus and aural fullness. It is more frequently unilateral than bilateral. Episodic vertigo is considered the most prominent symptom, with episodes typically lasting at least 20 minutes and resulting in significant patient morbidity. The diagnosis is primarily a clinical one, since there are no specific diagnostic tests for Meniere's disease. The disease is known to wax and wane, but eventually results in irreversible sensorineural hearing loss at all frequencies in the affected ear. While the pathogenesis of Meniere's disease has not been elucidated, one well-accepted mechanism involves the dysregulation of labyrinth fluid volume/ion balance resulting in endolymphatic hydrops (Shea, 1993). The increase in fluid volume and consequent increased labyrinth pressure may then be expressed as the Meniere's spectrum of symptoms.

There is no cure for Meniere's disease. Treatment tends to focus on relieving the vertigo symptoms, where it is hypothesized that reducing inner ear fluid volume will relieve the hydrops and associated clinical picture. It is for this reason that many subjects are initially started on low salt diets and diuretics (Barritt, 2008). A number of medical systemic treatments are also used to relieve Meniere's disease symptoms, including but not limited to antihistamines, anticholinergics, phenothiazines, benzodiazepines, and corticosteroids; however, these interventions are often inadequate in relieving the symptoms of Meniere's disease. A device that generates low-pressure pulses, the Meniett® device, is indicated for the symptomatic treatment of Meniere's disease. However, the device is not widely used and is not currently considered standard of care (Kim et al. 2005). Surgical decompression may be attempted in severe cases unresponsive to medical intervention, but surgical outcomes are frequently unsatisfactory. Finally, patients with unresponsive disease may undergo chemical or surgical neuroablation, resulting in symptom relief at the cost of destruction of the 8th cranial nerve. Thus, there continues to be an unmet medical need for therapies to address this debilitating disease.



# 1.1. Rationale for Safety Study

Two clinical studies have been conducted in the United States: a Phase 1b study and a Phase 2b study. The randomized, placebo-controlled, double-blind, multi-center Phase 2b study in 154 unilateral Meniere's disease patients demonstrated that a single IT administration of OTO-104 resulted in improvements in vertigo control. The completed and ongoing clinical studies have been either single-dose with a 3-month or 4-month follow-up period or a repeat-dose with 4 doses administered over one year. Because Meniere's disease is chronic and intermittent, the safety of repeat administration needs to be evaluated. This study was designed with a two injection design to look at repeat doses over the course of six months. Three months was chosen as the dose interval due to information gained during the follow-up period in regard to effect and safety in the completed Phase 1b and Phase 2b studies.

#### 2. OBJECTIVES

The objective is to assess the safety of repeat IT injections of 12 mg OTO-104 at 3-month intervals in an open-label study in subjects with unilateral Meniere's disease.

#### 3. OVERVIEW OF STUDY DESIGN

This is a 6-month, multicenter, Phase 3, open-label extension safety study in subjects with unilateral Meniere's disease. Subjects will receive 1 IT injection of 12 mg OTO-104 at 3-month intervals for a total of 2 injections. Safety data to be collected include adverse events, concomitant medications, otoscopy, vital signs, audiology, tympanometry, Columbia-Suicide Severity Rating Scale (C-SSRS) questionnaire and a Meniere's disease symptom questionnaire.

Once subjects meet all eligibility criteria, they will be enrolled and may receive up to 2 IT injections of OTO-104 at 3-month intervals. All subjects will remain on standard of care treatment for unilateral Meniere's disease. Subjects will return to the study sites at Month 3 for safety assessments and another IT injection of OTO-104. Safety assessments will be completed at the end of the study (Month 6) or upon early withdrawal from the study.

#### 4. STUDY POPULATION

#### 4.1. General Considerations

Up to 300 subjects will be enrolled at approximately 60-70 sites in the United States. Subjects will be enrolled only if they meet all of the inclusion criteria and none of the exclusion criteria

#### 4.2. Inclusion Criteria

Subjects enrolled in the study will have unilateral Meniere's disease as outlined by the American Academy of Otolaryngology - Head and Neck Surgery (AAO-HNS) Committee on Hearing and Equilibrium in 1995 (Committee on Hearing and Equilibrium, 1995).

To be eligible for this study, each of the following criteria must be satisfied with a "YES" answer (unless not applicable):

- 1. Subject is a male or female aged 18 years or older.
- 2. Subject has completed the Phase 2b (104-201102) or Phase 3 (104-201506) clinical study.
- 3. Female subjects of childbearing potential [i.e., not surgically sterile and/or not postmenopausal (12 months since last menstrual period and 45 years of age or older)] must have a negative urine pregnancy test before enrollment. Women of childbearing potential who are not abstinent from sex with male partners may be entered into the study if they are using and willing to continue to use highly effective or "double barrier" contraceptive precautions for the duration of the study (e.g., oral contraceptives, contraceptive implant or injection, intrauterine device, or "double barrier" methods including condom with diaphragm, male condom with cervical cap, male condom with spermicide, or diaphragm and spermicide).
- 4. Subject is willing to comply with the protocol and attend all study visits.
- 5. Subject is able to provide written informed consent, including agreement to privacy language either within the informed consent or in ancillary documents compliant with Health Insurance Portability and Accountability Act (HIPAA), before the initiation of any study-related procedures.

#### 4.3. Exclusion Criteria

To be eligible for this study, each of the following criteria must be satisfied with a "NO" answer: (unless not applicable):

- 1. Subject has an infection in the ear, sinuses, or upper respiratory system.
- 2. Subject is pregnant or lactating.
- 3. Subject has a history of immunodeficiency disease.
- 4. Subject has active or recent (<1 month prior to screening) middle ear disease, including but not limited to: chronic otitis media, acute otitis media, middle ear effusions, middle ear atelectasis, or cholesteatoma.

- 5. Subject has an abnormality of the tympanic membrane in the affected ear that would increase the risk associated with intratympanic injection including but not limited to a monomeric, atelectatic or atrophic tympanic membrane.
- Subject has a history of tympanostomy tubes that includes evidence of perforation or lack of closure.
- 7. Subject has a history of previous endolymphatic sac surgery.
- 8. Subject has a history of previous use of intratympanic gentamic in the affected ear.
- 9. Subject has history of drop attacks.
- 10. Subject has used systemic steroids within 1 month prior to Visit 1.
- 11. Subject has had intratympanic steroids within 1 month prior to Visit 1.
- 12. Subject has experienced an adverse reaction to intratympanic injection of steroids.
- 13. Subject has a hypersensitivity to dexamethasone or any of the excipients in OTO-104.
- 14. Subject has any other clinically significant illness or medical condition that, in the investigator's and the medical monitor's opinion, would prohibit the subject from participating in the study.
- 15. Subject has participated in a clinical trial within 30 days of Visit 1, not including the OTO-104 Phase 3 study (104-201506).

#### 5. RANDOMIZATION AND BLINDING

This study is an open-label study with all subjects receiving OTO-104; therefore, no randomization or blinding is required.

#### 5.1. Enrollment Procedures

#### 5.1.1. Assignment of Subject Identification Numbers

All subjects will retain the same unique subject identification number as the one assigned in clinical study 104-201102 or 104-201506 plus a 3-digit number to indicate which study the subject participated in previously. The subject identification number will be used to identify the subject throughout the study and will remain with the subject throughout the duration of the study. All subjects with a signed informed consent for the study, whether enrolled or not (screen failures, subject refusal, etc.), will be documented.

#### 6. DOSAGE AND ADMINISTRATION

# 6.1. Study Drug Administration

OTO-104 12 mg will be administered as a single, 0.2 mL intratympanic injection of 60 mg/mL OTO-104. The recommended injection procedure for intratympanic administration of OTO-104 in Meniere's disease subjects is as follows:

- 1. Place the subject in a recumbent position with the treated ear upwards. Anesthetize the tympanic membrane by covering the external surface of the posterior inferior quadrant with topical lidocaine/prilocaine cream (i.e., until the tympanic membrane is numb. If applicable, suction away the topical lidocaine/prilocaine cream.
- 2. Using the 1 mL syringe pre-loaded with OTO-104 and equipped with a 25 or 26 gauge needle, insert the needle through the tympanic membrane with the bevel facing in an inferoposterior direction to a depth of approximately 2-3 mm just inferior to the round window niche, and with firm but gentle pressure, inject 0.2 mL taking care not to insert the needle further than necessary. Use of this technique will minimize the possibility of OTO-104 adhering to the underside of the tympanic membrane. Do not incise the tympanic membrane to form a ventilation hole as this is not needed due to the small injection volume.

# 6.2. Compliance

OTO-104 will be administered by site personnel as a single, intratympanic injection at Visit 1 and 2 except when withheld due to potential safety concerns. Any deviations in administration will be documented in the source documents and the eCRF.

The site will maintain a log of all study drug dispensed and returned. Drug supplies for each subject will be inventoried and accounted for throughout the trial.

# 7. PRIOR, CONCOMITANT, AND SUBSEQUENT THERAPY

Use of all concomitant medications will be recorded in the subject's eCRF. This will include all symptomatic relief medications for Meniere's disease symptoms, prescription drugs, herbal products, vitamins, minerals, and over-the-counter medications taken within 30 days before enrollment, which will be considered prior therapy. Any concomitant medication deemed necessary for the welfare of the subject during the study may be given at the discretion of the Investigator except for those listed in Section 7.1. Any changes in concomitant medications will be recorded in the subject's eCRF.

# 7.1. Proscribed Therapy or Procedures During the Study Period

The following therapies are prohibited during the study:

- Systemic corticosteroids
- Immunosuppressive medications
- Phenol for use in anesthetizing the tympanic membrane
- Intratympanic injection other than that outlined in the current study
- Surgery for treatment of Meniere's disease
- Other investigational drug(s) or device(s)

Use of any of these proscribed therapies will be considered a protocol deviation.

# 7.2. Symptomatic Relief Medications

It is recognized that subjects may at times use certain medications for relief of symptoms related to Meniere's disease during the course of the study. Intermittent use of vestibular suppressants and anti-emetics is allowed as symptomatic relief medications. The use of gentamicin, corticosteroids or surgery at any time during the study will be considered a protocol deviation. Any changes reported by the subjects in concomitant medications should be recorded in the subject's eCRF.

#### 8. STUDY EVALUATIONS

# 8.1. Study Procedures by Visit

#### 8.1.1. Visit 1: Day 1 (Screening/Baseline/Dose No. 1)

The following assessments will be performed at Visit 1. For subjects enrolling directly (within 1 month) from Study 104-201506, the tympanometry, audiometry, otoscopy and C-SSRS assessment data collected at the final visit of Study 104-201506 will serve as the Baseline data for Visit 1.

The following assessments will be performed at Visit 1.

- Informed consent
- Confirm eligibility criteria
- Medical history
- Concomitant medications
- Vital signs
- Height and weight measurements
- Urine pregnancy test (for female subjects of childbearing potential only)
- Tympanometry
- Audiometry
- Otoscopy
- C-SSRS assessment: Baseline version or Since Last Visit version
- Meniere's symptom questionnaire
- Administer OTO-104 (all assessments in the above list must be conducted prior to OTO-104 administration)
- Adverse events (to be collected during or after OTO-104 administration)

## 8.1.2. Visit 2: Month 3 ( $\pm$ 2 weeks) (Follow Up and Dose No. 2)

The following assessments will be performed at Visit 2.

- Concomitant medications
- Vital signs
- Urine pregnancy test (for female subjects of childbearing potential only)
- Audiometry
- Tympanometry
- Otoscopy
- C-SSRS assessment, Since Last Visit version
- Meniere's symptom questionnaire
- Administer OTO-104 (all assessments in the above list must be conducted prior to OTO-104 administration)
- Adverse events (to be collected during or after OTO-104 administration)

## 8.1.3. Visit 3: Month 6 ( $\pm$ 2 weeks) (End of Study/Early Termination)

The following assessments will be performed at Visit 3.

- Concomitant medications
- Vital signs
- · Weight measurement
- Urine pregnancy test (for female subjects of childbearing potential only)
- Tympanometry
- Audiometry
- Otoscopy
- C-SSRS assessment, Since Last Visit version
- Meniere's symptom questionnaire
- Adverse events

#### 8.1.4. Unscheduled Visit

The following assessments will be performed at an unscheduled visit.

- Concomitant medications
- Vital signs
- · Tympanometry, as indicated
- Audiometry, as indicated
- Otoscopy
- C-SSRS assessment, Since Last Visit version

Adverse events

# 8.2. Safety Evaluations

Safety assessments include:

- Vital Signs, Height and Weight Measurements
- Tympanometry
- Audiometry
- Otoscopy
- C-SSRS Assessment
- Concomitant Medications
- Adverse events (see Section 9)

#### 8.2.1. Vital Sign, Height and Weight Measurements

Vital sign measurements (including systolic and diastolic blood pressure and pulse rate) will be collected at all study visits. Blood pressure and pulse rate will be measured after subjects have been seated for 5 minutes and while subjects are in a sitting position. Height and weight will be measured at Visit 1 and weight will be measured again at Visit 3.

# 8.2.2. Urine Pregnancy Test

A urine pregnancy test via dipstick will be conducted only on women of childbearing potential at all study visits. The urine pregnancy test must be conducted and confirmed negative prior to administration of OTO-104 at Study Visits 1 and 2.

#### 8.2.3. Tympanometry

Tympanometry assessments will be used to assess the mobility and compliance of the tympanic membrane, pressure and volume in the middle ear, and function of the tympanic membrane, ossicles and eustachian tube. Tympanograms will be completed in both ears at all study visits. Subjects wearing hearing aids should be instructed not to wear their hearing aids during the tympanometry assessment.

#### 8.2.4. Audiograms

Audiometric assessments will be used to assess hearing function in both ears. Audiograms should be conducted at 500, 1000, 2000, 4000 and 8000 Hz for both air and bone conduction at all study visits. Both air and bone conduction thresholds will be assessed. Pure tone averaging bone and air conduction testing will be done at 500, 1000, and 2000 Hz frequencies. Subjects wearing hearing aids should be instructed not to wear their hearing aids during the audiogram.

Audiometric assessments must be conducted in accordance with American-Speech-Language-Hearing Association Guidelines (ASHA, 2005). Equipment calibration must be current and documented. The audiometric assessments must be conducted by a licensed audiologist or a qualified assistant with appropriate training under the direct supervision of a licensed audiologist.

## 8.2.5. Otoscopy

Otoscopic exams will be used to assess the auditory canal, the appearance of the tympanic membrane, and the healing of the intratympanic injection site. Otoscopic examinations will be performed in both ears at all study visits during the study by the physician. Presence and size of tympanic membrane perforations will be recorded. Perforations of the tympanic membrane will be captured as adverse events (AEs) only if the perforation increases in size and does not resolve by the end of the study. Subjects wearing hearing aids should be instructed not to wear their hearing aids during the otoscopic exam.

#### 8.2.6. C-SSRS Assessment

The C-SSRS assessment will be administered at all study visits. The Since Last Visit version of the C-SSRS will be used for subjects enrolling from Study 104-201506 while the Baseline version will be used for all subjects enrolling from Study 104-201102. The Since Last Visit version of the C-SSRS will be used at all subsequent visits. Any subject with a positive score on the Baseline version or an appearance of any new suicidal ideation or suicide behavior since the Baseline version (whether administered in this study or Study 104-201506) should be referred to their primary care provider for follow-up.

If a subject has any post-Baseline C-SSRS score of 1-3 for Ideation (i.e., a "yes" answer to Questions 1, 2, or 3) or a "yes" response to the Non-Suicidal Self-Injurious Behavior question) and the score is higher than the Baseline C-SSRS score, then this assessment should be recorded as an adverse event (AE). This information is reported as indicated in Section 9.1. (Possible AE terms: Suicidal plans, Suicidal ideation, Suicidal tendency, Suicidal behavior, Suicidal intention, Suicidal depression, Active suicidal ideation, Passive suicidal ideation, Self-injurious behavior without suicidal intent).

If a subject has any post-Baseline C-SSRS score of 4 or 5 for Ideation (i.e., a "yes" answer to question 4 or 5) and/or any questions answered yes for Suicidal Behavior (with the exception of a "yes" response to the Non-Suicidal Self-Injurious Behavior question), and this was not observed at Baseline, then this assessment should be recorded as a serious adverse event (SAE). This information is reported as indicated in Section 9.2.2.

#### 8.3. Additional Evaluations

#### 8.3.1. Meniere's Symptom Questionnaire

The Meniere's symptom questionnaire is a set of questions that will be administered at Study Visits 1, 2, and 3. Each question has 5 possible responses: 1) No Vertigo/No Tinnitus/No Ear Fullness/No Hearing Difficulty (depending on the question administered), 2) Mild, 3) Moderate, 4) Severe, and 5) Extremely Severe. This assessment is considered an additional endpoint.

# 9. ADVERSE EVENT (AE) REPORTING

Timely, accurate, and complete reporting and analysis of safety information from clinical trials will be conducted in accordance with Good Clinical Practice.

All AEs, including SAEs reported or observed during or after dosing with the study drug will be recorded on the AE page of the eCRF for all enrolled subjects. Information to be collected includes description of event, date of onset, investigator-specified assessment of the severity and relationship to study drug, date of resolution of the event, seriousness, any required treatment or evaluations, and outcome. Adverse events resulting from concurrent illnesses, reactions to concurrent illnesses, reactions to concurrent medications, or progression of disease states must also be reported. Perforations of the tympanic membrane will be captured as AEs only if the perforation increases in size and does not resolve by the end of the study.

If the existing medical condition worsens at any time after application of study drug, it should be recorded as an AE.

#### 9.1. Adverse Event Classification Definitions

#### **Adverse Event:**

An AE is any unfavorable and unintended diagnosis, symptom, sign, syndrome or disease which occurs during the study, having been absent at baseline, or, if present at baseline, appears to worsen.

This includes any occurrence that is new in onset or aggravated in severity or frequency from the baseline condition, including abnormal results of diagnostic procedures and/or laboratory test abnormalities, which are considered AEs if they:

- result in discontinuation from the study
- require treatment or any other therapeutic intervention
- require further diagnostic evaluation (excluding a repetition of the same procedure to confirm the abnormality)
- are associated with clinical signs or symptoms judged by the investigator to have a significant clinical impact

#### **Serious Adverse Event (SAE):**

An SAE is defined as any untoward medical occurrence that:

- results in death,
- is life-threatening (Note: the term "life-threatening" refers to an event in which the subject was at risk of death at the time of the event rather than to an event which hypothetically might have caused death if it were more severe.),
- requires in-patient hospitalization or prolongation of existing hospitalization,
- results in persistent or significant disability/incapacity, or
- is a congenital anomaly/birth defect.

Medical and scientific judgment should be exercised in deciding whether expedited reporting is appropriate in other situations, such as important medical events that may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes listed in the above definition. These events should be considered serious.

#### 9.1.1. Assessment of Severity

The investigator will assess the intensity of the AE and rate the AE as mild, moderate, or severe using the following criteria:

<u>Grade 1 - Mild:</u> These events are easily tolerated, require minimal or no treatment, and do not interfere with the subject's daily activities.

<u>Grade 2 – Moderate:</u> These events cause sufficient discomfort to interfere with daily activity and/or require a simple dose of medication, e.g., analgesics or anti-emetics.

<u>Grade 3 – Severe:</u> These events incapacitate and prevent usual activity or require complex medication/treatment or hospitalization.

<u>Grade 4 – Life Threatening:</u> These events are those for which the subject was at risk of death at the time of the event rather than an event which hypothetically might have caused death if it were more severe.

<u>Grade 5 – Death:</u> The event resulted in the death of the subject.

Changes in the severity of an AE should be documented to allow for an assessment of the duration of the event at each level of intensity to be performed.

#### 9.1.2. Assessment of Causality

The investigator's assessment of an AE's relationship to study drug will be part of the documentation process, but will not be a factor in determining what is or is not reported in the study.

The investigator will assess the relationship or association of the study drug in causing or contributing to the AE, which will be characterized using the following classification and criteria:

<u>Definite</u>: Adverse events that, after careful medical evaluation, are considered definitely related to the study drug; other conditions (concurrent illness, progression/expression of disease state, or concurrent medication reaction) do not appear to explain the event.

<u>Probable</u>: Adverse events that, after careful medical evaluation, are considered with a high degree of certainty to be related to the study drug. The following characteristics will apply:

- a reasonable temporal relationship exists between the event and exposure to the study drug, and
- the event is a known reaction to the study drug that cannot be explained by an alternative cause commonly occurring in the population/individual, or
- the event is not a known reaction to the study drug but cannot be reasonably explained by an alternative cause.

<u>Possible</u>: Adverse events that, after careful medical evaluation, do not meet the criteria for a definite or probable relationship to the study drug, but for which a connection cannot be ruled out with certainty. The following characteristics will apply:

- the event occurs after exposure to the study drug, and
- there is a reasonable temporal relationship to the application, but the event is not a known reaction to the study drug and could be explained by a commonly occurring alternative cause, or
- in the absence of a reasonable temporal relationship, the event cannot be explained by an alternative cause.

Not related: Adverse events in this category will have either of the following characteristics:

• the event does not have a reasonable temporal relationship to study drug administration and/or can be explained by a commonly occurring alternative cause.

## 9.1.3. Follow up of Adverse Events

The investigator will follow a non-serious AE until resolution, stabilization, or the End of Study Visit. The investigator will follow an SAE (regardless of relationship to study drug) until the event resolves, stabilizes, or becomes non-serious. All AEs identified on the last scheduled contact must be recorded on the AE page of the eCRF and the current status (ongoing or resolved) will be noted. In addition, SAEs will be reported to Product Safety according to the reporting guidelines identified in Section 9.2.2.

# 9.2. Monitoring of Adverse Events

#### 9.2.1. All Adverse Events

All AEs will be analyzed for safety. Those meeting the definition of SAE must be reported using the SAE Form. Subjects should voluntarily report any AEs or report AEs in response to general, non-directed questioning (e.g., "How has your health been since the last visit?"). For each AE volunteered by the subject, the investigator should obtain all the information required to complete the AE page of the eCRF, in accordance with the guidelines that accompany it.

All AEs, regardless of seriousness, severity, or presumed relationship to study therapy, must be recorded using medical terminology in the source document and on the eCRF. Whenever possible, diagnoses should be given when signs and symptoms are due to a common etiology (e.g., cough, runny nose, sneezing, sore throat, and head congestion should be reported as "upper respiratory infection"). Investigators must record on the eCRF their opinion concerning the relationship of the AE to study therapy. All measures required for AE management must be recorded in the source document and reported according to sponsor instructions.

Any non-serious AE that occurs after the dose of study drug must be reported in detail on the appropriate eCRF page and followed until resolution, stabilization, or the End of Study Visit. The description of the AE will include description of event, date of onset, date of resolution, investigator assessment of severity and relationship to study drug, seriousness, any required treatment or evaluations, and outcome.

The sponsor assumes responsibility for appropriate reporting of AEs to the regulatory authorities. The sponsor will also report to the investigators all serious AEs that are unlisted and associated with the use of the drug. The investigators must report these events to the appropriate Institutional Review Board (IRB) in accordance with local regulations.

#### 9.2.2. Serious Adverse Events

All SAEs occurring during clinical trials must be reported within 24 hours to Product Safety.

The cause of death of a subject in a clinical trial, whether the event is expected or associated with the investigational agent, is an SAE.

The initial report of an SAE may be made by telephone, e-mail or facsimile (fax). The investigator must provide the minimal information: i.e., protocol number, subject's initials and date of birth, subject number or medication code number, nature of the AE and investigator's attribution.

All oral reports of an SAE must be confirmed within 24 hours by a written, more detailed report and signed by the investigator. For this purpose, the sponsor will provide the investigator with the Serious Adverse Event Form for Clinical Trials.

All SAEs that have not resolved by the end of the study, or that have not resolved upon discontinuation of the subject's participation in the study, must be followed until either:

- the event resolves,
- the event stabilizes, or
- the event becomes non-serious

The investigator should report any follow-up information as it becomes available.

#### 9.2.3. Pregnancies

Pregnancies occurring after the first dose of investigational product and during participation of the study are considered immediately reportable events. While not considered a SAE unless a serious criterion is met, pregnancies occurring in subjects enrolled on the study must be reported and followed to outcome. The investigator should complete the pregnancy report eCRF within one working day of knowledge of the pregnancy. Following delivery or termination of pregnancy, the follow-up pregnancy report form should be completed on the pregnancy CRF. Spontaneous abortions should always be reported as SAEs. Follow-up information regarding the outcome of the pregnancy and any postnatal sequelae in the infant will be required.

# 9.3. Contacting Sponsor Regarding Safety

Any AE considered serious by the investigator, or that meets the SAE criteria stated in this protocol, must be reported to Product Safety within 24 hours from the time that study site personnel first learns of the event. The study site must enter the SAE into the EDC system.

Source documents will be requested from the study sites for SAEs and should be provided to Product Safety. If the subject is hospitalized during the study, a copy of the hospital discharge summary should be provided to the Product Safety as soon as it becomes available.

# 10. SUBJECT COMPLETION

# 10.1. Completion

Subjects who withdraw from further administration of study drug or who withdraw their consent to be followed or are lost-to-follow-up before completion of Visit 3 (Month 6) will not be considered to have completed the study.

#### 10.2. Withdrawal

All subjects have the right to withdraw from study drug administration and/or study evaluations at any time, for any reason, without prejudice; nonetheless, investigators should attempt to encourage subjects to complete the protocol even if the subject has withdrawn from study drug so that continued observation and follow-up measurements may be obtained. The investigator may discontinue a subject's participation in the study at his/her discretion for reasons including, but not limited to, the following:

- 1. Subject experiences a serious or intolerable AE that, in the opinion of the investigator, requires withdrawal from the study.
- 2. Subject is in violation of the protocol.
- Subject develops a condition during the course of the study that makes it unwise to continue with the trial.
- 4. Subject requires a medication that is prohibited by the protocol.
- 5. Subject requests an early discontinuation for any reason.

At any point, the investigator may discontinue the subject's study participation at his/her discretion and ensure the subject receives appropriate medical care; the investigator may also consult the medical monitor to discuss out-of-range test results.

#### 10.2.1. Handling of Withdrawals

Subjects will be free to withdraw from further study drug administration and further follow-up the study at any time. Subject participation in the study may be stopped at any time at the discretion of the investigator or at the request of the sponsor.

Whenever possible, all subjects who withdraw from further study drug administration should be encouraged to remain on-study for further follow-up through the subject last scheduled visit. However, should a request for early withdrawal from the study with no further follow-up be made, the subject should be encouraged to return to the study site for a last follow up visit and undergo all end of study/early termination assessments.

When a subject withdraws from further administration of study drug or the study prior to completing Visit 3 (Month 6), the reason for withdrawal is to be documented on the eCRFs and in the source document.

# 10.2.2. Replacements

Subjects who discontinue participation in the study for any reason after dosing will not be replaced.

#### 11. STATISTICAL METHODS

The emphasis of the analysis will be with respect to description and estimation rather than hypothesis testing. The following statistical sections describe the general analytic methods to be implemented to assess the overall study objectives. More detailed descriptions of the methodology will be provided in the Statistical Analysis Plan (SAP).

# 11.1. Sample Size

It is expected that up to 300 subjects from Phase 2b (104-201102) or Phase 3 (104-201506) clinical trials will be enrolled into this study. The sample size was not based on any power calculation.

# 11.2. Analysis Sets

The following definitions will be used to derive the analysis sets for this study.

<u>Safety Analysis Set</u>: The safety analysis set will include all subjects who receive at least one dose of study drug.

# 11.3. Description of Subgroups to be Analyzed

Key safety data will be described for the following subgroups using the safety analysis set:

- Subject Demographics
  - Gender

Additional demographic and baseline characteristic subgroups will be considered and identified in detail in the SAP.

# 11.4. Subject Demographics, Baseline Disease Status, and Disposition

Descriptive statistics for subject demographics, baseline disease status, and subject disposition will be provided. If feasible, a Kaplan-Meier plot of time-to-study withdrawal will also be estimated. Protocol deviations will be analyzed by aggregate summary and/or line listings if the number of deviations is small.

# 11.5. Efficacy Evaluations

Not applicable

# 11.6. General Analytic Methods

The primary analytic approach for this trial will be descriptive. Summary statistics will be calculated and where relevant, 95% confidence intervals presented. Details of the analysis will be described in the SAP.

# 11.7. Safety Evaluations

Safety evaluations include:

- Vital Signs, Height and Weight Measurements
- Tympanometry
- Audiometry
- Otoscopy
- C-SSRS Assessment
- Concomitant Medications
- Adverse events

#### 11.7.1. Adverse Events

Version 18.1 of Medical Dictionary for Regulatory Activities (MedDRA) will be used to code all AEs.

The primary analysis of AEs will consider only treatment emergent AEs (TEAEs), events occurring for the first time, or worsening during or after the first dose of study drug. Subject incidence of TEAEs and SAEs will be tabulated by preferred terms and system organ class. These analyses may also be tabulated by visit, time of onset and/or cumulative exposure. In addition, severity and relationship to study drug will also be presented. Adverse events will be presented by descending order of frequency in MedDRA system organ class and preferred term.

Subgroup analyses of AEs by gender will be examined. Listings of all SAEs, AEs leading to study withdrawal, and deaths on-study will also be included. Duration and outcome of each AE will be reported in subject listings.

#### **11.7.2.** Vital Signs

The analysis of vital signs will include descriptive statistics for the change from baseline to each post-baseline visit where vital signs are collected. The change from baseline to the worst post-baseline value (increase/decrease) may also be examined. Weight measurements for baseline and post-baseline visits will be tabulated as will height measurements for baseline.

#### 11.7.3. Otoscopic Examinations

Observations recorded during the conduct of otoscopic exams will be descriptive. The number and percent of subjects presenting with each otoscopic classification will be provided by study visit using shift tables where appropriate. Data will be tabulated separately for the treated and untreated ear.

#### 11.7.4. Audiometry Assessments

Descriptive summary statistics and/or shift tables for audiometric assessments of air and bone conduction thresholds at each frequency will be provided by study visit. In addition, the pure tone average (PTA) and bone conduction average (BCA) will be calculated as the average air or bone conduction threshold for frequencies of 500, 1000, and 2000.

Air-Bone Gap assessments at each frequency and study visit will be tabulated as the proportion of subjects with air minus bone conduction thresholds of

- < 10 dB or</p>
- > 10 dB.

All audiometry assessments will be tabulated separately for the treated and untreated ear.

## 11.7.5. Tympanometry

Shift tables representing the proportion of subjects with changes in their tympanogram from baseline to each post-baseline study visit will be calculated. Tympanogram changes will include both the type of tympanogram (A, B-small volume and/or normal, B-large volume, or C).

#### 11.7.6. Concomitant Medications

Concomitant medications will be coded by WHO Drug and will be tabulated by drug class and preferred drug name.

#### 11.7.7. C-SSRS

The C-SSRS will be administered at each visit using the appropriate version i.e. Baseline or Since Last Visit. Analysis of this scale will be performed on the Safety Analysis Set.

#### 11.7.7.1. C-SSRS: Baseline Version

The C-SSRS assessment will be administered at all study visits. The Since Last Visit version of the C-SSRS will be used for subjects enrolling directly (within 1 month) from Study 104-201506 while the Baseline version will be used for all other subjects. The Since Last Visit version of the C-SSRS will be used at all subsequent visits. The Baseline version of the scale captures both suicide ideation and suicide behavior (lifetime). There are 5 suicidal ideation questions, each captured as yes/no for the subject's lifetime. Additionally a sixth suicidal ideation variable will be created to indicate if there was any ideation, regardless of type. There are 4 suicidal behavior questions, each captured as yes/no for the subject's lifetime. A fifth suicidal behavior variable will be created to capture if there was any suicidal behavior regardless of type. An additional question asks if suicidal behavior is present during the visit. All suicidal ideation and behavioral variables as outlined here will be tabulated overall and by treatment group. All C-SSRS data will be included in data listings. There is no inclusion or exclusion criterion associated with the Baseline C-SSRS score.

#### 11.7.7.2. C-SSRS: Since Last Visit Version

The Since Last Visit version of the C-SSRS will be administered at each study visit including Visit 1 or after Visit 1 depending on whether the subject was a participant from Study 104-

201102 or 104-201506. The same overall individual variables for suicidal ideation and behavior will be assessed as in the Baseline version. In addition, overall suicidality (yes/no) will be defined as any subject having any suicidal ideation or behavior since the last visit. All suicidal ideation and behavior variables will be tabulated overall and by treatment group for each study visit. All C-SSRS data will be included in data listings.

#### 11.8. Other Evaluations

Additional endpoints include:

• Meniere's symptom questionnaire

#### 11.8.1. Meniere's Symptom Questionnaire

Descriptive summary statistics denoting the change from baseline and/or shift tables for the vertigo, tinnitus, aural fullness and subjective hearing will be provided. For the Global Meniere's Disease question, not measured at baseline, summary statistics for each visit will be provided.

# 11.9. Handling of Missing Data, Subject Withdrawals, and Treatment Failures

Every effort will be made to follow subjects for study observation and encourage compliance with study measurements to minimize the amount of missing data.

Except for partial dates, safety data will not be imputed. The imputation algorithm for partial dates will be defined in the SAP.

# 11.10. Interim Analyses

There are no formal interim analyses planned. Review of safety data will be conducted as described in Section 14.7; however, the review of such data is not intended to impact the study conduct unless there are safety concerns. As such, it is expected that the trial will continue to its scheduled completion barring any unexpected safety issues.

#### 12. STUDY DRUG INFORMATION

# 12.1. Physical Description of Study Drug(s)

The investigational drug product administered to subjects in this study will be OTO-104. The OTO-104 final product suspension for dosing will be prepared from two separate components, OTO-104 Diluent (one vial needed) and OTO-104 Active (one vial needed). An appropriate volume of OTO-104 Diluent will be withdrawn and delivered into the OTO-104 Active vial to achieve a visually homogeneous suspension of a target drug concentration of 60 mg/mL.

The product will be supplies as a kit containing one vial of OTO-104 Active and one vial of OTO-104 Diluent.

## 12.2. Directions for Use

OTO-104 is to be prepared in a clean location with a room temperature preferably at or below 23°C (73°F). Please refer to the Pharmacy Manual for detailed study drug preparation instructions.

# 12.3. Packaging and Labeling

#### 12.3.1. Packaging

All study drug kits will be labeled with information that will meet the applicable regulatory requirements.

#### 12.3.2. Labels and Labeling Instructions

A label will be affixed to each kit box, OTO-104 Active and OTO-104 Diluent vials indicating contents and storage instructions.

# 12.4. Management of Clinical Supplies

The clinical supplies will be managed by the CRO. The Sponsor will create shipment requests that will be generated on inventory thresholds that are set for each site. A shipment request will be generated and sent to the clinical supplies vendor. Upon shipment and receipt of the clinical trial material, the site personnel will acknowledge the shipment and identify any damaged, missing, or unusable kits so they will not be dispensed.

## 12.4.1. Storage of Kits

All kits will be stored at  $-20^{\circ}$ C ( $\pm 5^{\circ}$ C), with allowable temperature excursions as high as  $25^{\circ}$ C for up to 72 hours. All temperature excursions of the study drug must be documented in the study drug accountability log. Any excursions within the allowable temperature range and conditions should be documented, but the study drug is still acceptable for use and dispensing to subjects. If any excursions are outside of these conditions, the study drug should not be used to treat subjects. If this occurs, the study drug should immediately be quarantined and removed from inventory.

# 12.5. Drug Accountability

It is the responsibility of the clinical investigator to ensure that all study drug received at the site will be inventoried and accounted for throughout the study and the result recorded on the drug accountability form maintained in the Pharmacy Manual. The must return all original containers, whether empty or containing study drug, when instructed by the study monitor to return. Study drug returned by the clinical site staff will be stored and disposed of according to the sponsor's instructions. Drug accountability will be verified by the sponsor's study monitor during on-site monitoring visits. Study drug will be stored in a limited access area or in a locked cabinet under appropriate environmental conditions.

The investigator agrees not to supply the study drug to any person other than sub-investigators, designated staff and the subjects participating in the study. Study drug may not be relabeled or reassigned for use by other subjects except under special circumstances approved by Otonomy.

The investigator will retain and store all original containers returned by the clinical site staff until these containers are inventoried by the study monitor. Unless otherwise instructed by the sponsor, the investigator agrees at the end of the study to return all original containers, whether empty or containing study drug, to the sponsor as instructed by the study manager. The investigator agrees to neither dispense the study drug from, nor store it at, any site other than the study sites agreed upon with the sponsor.

The sponsor will ensure proper disposition of original containers empty or full with returned or unused study drug. Appropriate documentation will be maintained. Permission may be granted for local disposition, with supporting documentation.

#### 13. ETHICAL ASPECTS

# 13.1. Investigator Responsibilities

The investigator is responsible for ensuring that the clinical study is performed in accordance with the protocol, the Declaration of Helsinki, as well as with the Note for Guidance on Good Clinical Practice (ICH/135/95), and applicable regulatory requirements. These documents set forth that the informed consent of the subjects is an essential precondition for participation in the clinical study.

# 13.2. Institutional Review Board (IRB)

This trial will be undertaken only after full approval of the protocol and addenda has been obtained from a designated IRB and the sponsor has received a copy of this approval.

The IRB must be informed of all subsequent protocol amendments issued by the sponsor.

Reports on, and reviews of, the trial and its progress will be submitted to the IRB by the investigator at intervals stipulated in their guidelines.

#### 13.3. Informed Consent

Each subject must give written consent (and sign other locally required documents) according to local requirements after the nature of the study has been fully explained. The consent form must be signed prior to performance of any study-related activity. The consent form that is used must be approved both by the sponsor and by the reviewing IRB. The informed consent should be in accordance with the current revision of the Declaration of Helsinki, current International Conference on Harmonization (ICH) Good Clinical Practice (GCP) guidelines, and Otonomy policy.

The investigator must explain to potential subjects the aims, methods, reasonably anticipated benefits and potential hazards of the trial and any discomfort it may entail. Subjects will be informed that they are free not to participate in the trial and that they may withdraw consent to participate at any time. They will be told which alternative treatments are available if they refuse to take part, and that such refusal will not prejudice future treatment. Finally, they will be told that their records may be examined by competent authorities and authorized persons, but that personal information will be treated as strictly confidential and will not be publicly available. Subjects must be given the opportunity to ask questions. After this explanation and before entry

into the trial, consent should be appropriately recorded by means of the subject's dated signature. If a subject is unable to read, an impartial witness must be present during the entire informed consent discussion. The signature of the impartial witness will certify the subject's consent. The subject should receive a signed and dated copy of the informed consent form.

# 14. ADMINISTRATIVE REQUIREMENTS

#### 14.1. Protocol Modifications

All protocol amendments must be issued by the sponsor, signed and dated by the investigator, and should not be implemented without prior IRB approval, except where necessary to eliminate immediate hazards to the subjects or when the change(s) involves only logistical or administrative aspects of the trial (e.g., change in monitor, change of telephone number). Responsibilities for reporting protocol amendments to any Regulatory Authority (if applicable) and/or IRB are further described in the Ethical Aspects section of the protocol.

In situations requiring a departure from the protocol, the investigator or other physician in attendance will contact the site manager, Medical Monitor or other appropriate sponsor representative by fax, email or telephone (see Sponsor Contact Information page). If possible, this contact will be made before implementing any departure from protocol. In all cases, contact with the sponsor must be made as soon as possible in order to discuss the situation and agree on an appropriate course of action. The eCRF and source document will describe any departure from the protocol and the circumstances requiring it.

# 14.2. Regulatory Documentation

Documents that must be provided to the sponsor prior to study drug shipment are as follows:

- Up-to-date curriculum vitae for each investigator and sub-investigator.
- Signed and dated Investigator Agreement.
- Applicable local regulatory documentation
- A copy of the formal written notification to the investigator regarding approval of the
  protocol by an IRB that is in compliance with regulatory guidelines. The written
  notification is to be signed by the chairman or authorized designee and must identify
  the specific protocol. In cases where an IRB member has a known conflict of
  interest, abstention of that individual from voting should be documented; an
  investigator (or sub-investigator) may be a member of the IRB, but may not vote on
  any research in which he or she is involved.
- Financial disclosure documentation for each investigator and sub-investigator.
- Name and address of the IRB with a statement that it is organized and operates
  according to GCP and the applicable laws and regulations, and a current list of the
  IRB members. The IRB Attestation form can be used to capture this information.

- A copy of the IRB approved informed consent form and other adjunctive materials (e.g., advertising) to be used in the study, including written documentation of IRB approval of these items.
- Required financial agreement.

In addition to the documents required prior to the study, other documentation may be required during the course of the study.

# 14.3. Subject Identification Register

The investigator agrees to complete a subject identification register, which will be used for the purpose of long-term follow-up, if needed. This form will be treated as confidential, and will be filed by the investigator in the Trial Site File. Otherwise, all reports and communications relating to the study will identify subjects by initials and assigned number only.

#### 14.4. Record Retention

In compliance with the ICH/GCP guidelines the investigator/institution will maintain all eCRFs and all source documents that support the data collected from each subject, and all trial documents as specified in Essential Documents for the Conduct of a Clinical Trial and as specified by the applicable regulatory requirement(s). The investigator/institution will take measures to prevent accidental or premature destruction of these documents. Essential documents must be retained until at least two years after the last approval of a marketing application in an ICH region or at least two years have elapsed since the formal discontinuation of clinical development of the investigational product. These documents will be retained for a longer period if required by the applicable regulatory requirements or by an agreement with the sponsor. It is the responsibility of the sponsor to inform the investigator/institution as to when these documents no longer need to be retained. If the responsible investigator retires, relocates, or for other reasons withdraws from the responsibility of keeping the study records, custody must be transferred to a person who will accept the responsibility. The sponsor must be notified in writing of the name and address of the new custodian.

# 14.5. Electronic Case Report Form

Electronic Case Report Forms (eCRFs) will be completed for each subject. Access for data entry will be provided to appropriate site staff members. All data must be entered into the eCRFs in English and signed and dated electronically by the investigator.

The eCRFs should be completed by investigator site staff at the time of the subject's visit, with the exception of results of tests performed outside the investigator's office, so that they always reflect the latest observations on the subjects participating in the trial.

As the site staff enters data, discrepancies will be automatically generated within the Electronic Data Capture (EDC) system for the site staff to resolve immediately. In addition, as a result of data review by the Sponsor or designee, manual queries will be raised electronically in the EDC system. Queries may also be raised as a result of source data verification by the clinical monitor. All corrections will be made within the EDC system by the investigator or other authorized study site personnel. The clinical monitor and data management teams will ensure appropriate

resolution of queries. The investigator must authorize changes to the recorded safety and efficacy data.

#### 14.6. Termination

An initiative for center closure or trial termination can be taken at any time either by the sponsor or by the investigator, provided there is reasonable cause and sufficient notice is given in advance of the intended termination. Reasons for such action taken by the sponsor include, but are not limited to:

- Successful completion of the trial at the center
- The maximum number of eligible subjects for the trial has been enrolled
- Failure of the investigator to comply with the protocol, the sponsor's procedures, or GCP guidelines
- Safety concerns
- Inadequate recruitment of subjects by the investigator
- Business reasons

# 14.7. Data and Safety Monitoring Plan

The sponsor shall promptly review all information relevant to the safety of the drug obtained or otherwise received from foreign or domestic sources, including information derived from this clinical study and any other clinical study conducted with OTO-104. In order to comply with this, the sponsor and CRO medical personnel will have the ability to review safety information as it is entered and verified in the electronic data capture system (Section 14.5). Depending on the enrollment rate, all AEs in the ear and labyrinth disorders SOC will be reviewed at least every other month. In addition, reasons for study discontinuation will be reviewed to see if any trends in study discontinuation are identified.

Investigators are instructed to contact the Product Safety within 24 hours following the identification of a SAE (Section 9.2.2). All SAEs will be reviewed by the sponsor and CRO medical personnel within 1-2 days after receipt whether or not the event was considered associated with study drug. The sponsor assumes responsibility for appropriate reporting to the regulatory authorities. The investigator assumes responsibility for reporting events to the IRB in accordance with the IRB requirements. All SAE's will be part of the CRO medical personnel/sponsor safety review.

If, through this ongoing review, the sponsor determines that OTO-104 presents an unreasonable and significant risk to subjects, the sponsor shall take appropriate steps to suspend or discontinue the study and notify regulatory authorities, investigators and IRBs as appropriate.

# 14.8. Monitoring

The sponsor or its representatives will perform on-site monitoring visits as frequently as necessary based on site activity to review protocol compliance, compare eCRFs with individual subject's medical records and clinic charts, and ensure that the study is being conducted according to pertinent regulatory requirements. The dates of the visits will be recorded by the

monitor in a trial center visit log to be kept at the site. The first post-initiation visit will usually be made as soon as possible after enrollment has begun. At these visits, the monitor will compare the data entered onto the eCRFs with the hospital or clinic records (source documents). The review of medical records will be performed in a manner that ensures subject confidentiality is maintained. At a minimum, source documentation must be available to substantiate proper informed consent procedures, adherence to protocol procedures, adequate reporting and follow-up of AEs, administration of concomitant medication, drug receipt/dispensing/return records, and study drug administration information. Specific items required as source documents will be reviewed with the investigator prior to the study. Findings from this review of eCRFs and source documents will be discussed with the investigator. The sponsor expects that, during monitoring visits, the investigator (and as appropriate, the study coordinator) will be available, the source documentation will be available, and a suitable environment will be provided for review of study-related documents.

# 14.9. Data Quality Assurance

Steps to be taken to assure the accuracy and reliability of data include the selection of qualified investigators and appropriate study centers, review of protocol procedures with the investigator and associated personnel prior to study initiation, and periodic monitoring visits by the sponsor or its representatives. Case report forms will be reviewed for accuracy and completeness in the EDC system database by the sponsor or its representatives during and after on-site monitoring visits, and any discrepancies will be resolved with the investigator or designees, as appropriate, and documented in the EDC system.

#### 14.10. On-Site Audits

Representatives of the sponsor's Quality Assurance department may visit the site to carry out an audit of the study in compliance with regulatory guidelines and company policy. Such audits will require access to all study records, including source documents, for inspection and comparison with the eCRFs. Subject privacy must, however, be respected. Sufficient prior notice will be provided to allow the investigator to prepare properly for the audit.

Similar auditing procedures may also be conducted by agents of any regulatory body reviewing the results of this study in support of a Licensing Application. The investigator should immediately notify the sponsor if they have been contacted by a regulatory agency concerning an upcoming inspection.

#### 14.11. Use of Information and Publication

All information concerning OTO-104, Otonomy operations, patent application, formulas, manufacturing processes, basic scientific data, and formulation information, supplied by the sponsor to the investigator and not previously published, is considered confidential and remains the sole property of Otonomy. The investigator agrees to use this information only to accomplish this study and will not use it for other purposes without the sponsor's written consent.

The investigator understands that the information developed in the clinical study will be used by Otonomy in connection with the continued development of OTO-104, and thus may be disclosed as required to other clinical investigators or government regulatory agencies. To permit the

information derived from the clinical studies to be used, the investigator is obligated to provide the sponsor with all data obtained in the study.

Any publication or other public presentation of results from this study requires prior review and written approval of Otonomy. Draft abstracts, manuscripts, and materials for presentation at scientific meetings should be provided to the sponsor at least 30 working days prior to abstract or other relevant submission deadlines. Authorship of publications resulting from this study will be based on generally accepted criteria for major medical journals.

## 15. LIST OF REFERENCES

American Speech-Language-Hearing Association. (2005). Guidelines for manual pure-tone threshold audiometry [Guidelines]. Available from www.asha.org/policy. - See more at: http://www.asha.org/policy/GL2005-00014.htm#sthash.0Xg5whCS.dpuf

Barritt L. Meniere's Disease. XPharm 2008 (1-6).

Committee on Hearing and Equilibrium. Committee on Hearing and Equilibrium guidelines for the diagnosis and evaluation of therapy in Meniere's disease. *Oto-laryngol Head Neck Surg.* 1995; 113(3):181-185.

Kim HH, Wiet RJ, Batista RA. Trends in the diagnosis and management of Meniere's disease: results of a survey. *Otolaryngol Head Neck Surg.* 2005; 132:722-6.

Shea JJ: Classification of Meniere's Disease. Am J Otol 1993: 14:224-229.